CLINICAL TRIAL: NCT05646004
Title: An Open Single-arm Clinical Investigation to Evaluate the Clinical Safety and Effectiveness of 621
Brief Title: 621 Real World Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 621P-BER-401-21
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Senile Cataract
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 621 (Experimental)
  Interventions: Device: Cataract surgery

INTERVENTIONS:
Device: Cataract surgery — Implantation of 621 lens

SUMMARY:
This study is evaluating the clinical safety and effectiveness of 621, after cataract surgery.

ELIGIBILITY:
Inclusion:

1. Age ≥ 18 years old;
2. Patient with clinically significant cataract with planned phacoemulsification cataract extraction and implantation of IOL into the capsular bag;
3. Preoperative corneal astigmatism ≤ 1.00D;
4. Patient is willing and capable of providing informed consent;
5. Patient is willing and capable of complying with visits and procedures as defined by this protocol.

Exclusion:

1. Preoperative best corrected visual acuity > 4.7 or ≤ 0.3 logMAR;
2. Corneal endothelial cell count less than 2000 cell/mm2;
3. Age under 18 years old;
4. Pregnant and lactating women;
5. Patients who attend other drug or medical device study;
6. Ocular disorder that could potentially cause a clinically significant future visual acuity loss;
7. Anterior segment pathology (e.g. chronic uveitis, iritis, aniridia, rubeosis iridis, anterior membrane dystrophies, poor pupil dilation, etc.)
8. Abnormal corneal finding (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism, clinically significant corneal membrane dystrophies);
9. Any condition in the study eye that could affect IOL stability (e.g. pseudo-exfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc;
10. Any acute infection (acute ocular disease, external/internal infection, systemic infection);
11. History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy, amblyopia, strabismus, microphthalmia, aniridia, epiretinal membrane etc.) in the study eye that could alter or limit final postoperative visual prognosis;
12. Any previous intraocular and corneal surgery ;
13. Uncontrolled glaucoma or IOP higher than 24mmHg under ocular hypertension treatment;
14. Current systemic or ocular pharmacotherapy that effects patients' vision;
15. Current pathology or condition that could be a risk for the patient according to the investigator opinion;
16. Patients unable to meet the limitations of the protocol or likely of non-cooperation during the clinical investigation;
17. Patients whose freedom is impaired by administrative or legal order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity (CDVA) | 6 months
  measurement of CDVA after IOL implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Boao Lecheng Aier Eye Hospital, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided